CLINICAL TRIAL: NCT01118481
Title: ADenosine Vasodilator Independent Stenosis Evaluation Study (ADVISE)
Brief Title: Vasodilator Free Measure of Fractional Flow Reserve
Acronym: ADVISE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Hospital San Carlos, Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 1428
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Stenosis
Keywords: Coronary stenosis; Wave intensity analysis; Instantaneous Flow Reserve; iFR; Fractional Flow Reserve
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pressure and flow velocity
- Pressure only

SUMMARY:
Narrowing of coronary arteries interferes with blood flow and can cause chest pain. Cardiologists sometimes quantify the extent of the narrowing by measuring the fractional flow reserve (the ratio of the pressure in the aorta to the pressure downstream of the narrowing under conditions of maximal flow). We propose a new technique based on principles of wave intensity analysis (WIA) to better assess coronary stenosis and the significance of the narrowing without the need for administration of vasodilator agents such as adenosine. This would simplify assessment and improve our ability to advise patients whether stent treatment will help their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary stenosis

Exclusion Criteria:

* Patient's with cardiac pacemakers, valvular heart disease, and chronic renal failure
* Unable to consent
* Contraindications to adenosine
* Contraindications to cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary stenosis without exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Correlation and descriptive characteristics between adenosine free measure of stenosis severity and FFR | Study end

CONTACTS AND LOCATIONS:
Overall Officials: Justin E Davies, BSc, MBBS, MRCP, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Sen S, Asrress KN, Nijjer S, Petraco R, Malik IS, Foale RA, Mikhail GW, Foin N, Broyd C, Hadjiloizou N, Sethi A, Al-Bustami M, Hackett D, Khan MA, Khawaja MZ, Baker CS, Bellamy M, Parker KH, Hughes AD, Francis DP, Mayet J, Di Mario C, Escaned J, Redwood S, Davies JE. Diagnostic classification of the instantaneous wave-free ratio is equivalent to fractional flow reserve and is not improved with adenosine administration. Results of CLARIFY (Classification Accuracy of Pressure-Only Ratios Against Indices Using Flow Study). J Am Coll Cardiol. 2013 Apr 2;61(13):1409-20. doi: 10.1016/j.jacc.2013.01.034. PMID 23500218
- [Derived] Sen S, Escaned J, Malik IS, Mikhail GW, Foale RA, Mila R, Tarkin J, Petraco R, Broyd C, Jabbour R, Sethi A, Baker CS, Bellamy M, Al-Bustami M, Hackett D, Khan M, Lefroy D, Parker KH, Hughes AD, Francis DP, Di Mario C, Mayet J, Davies JE. Development and validation of a new adenosine-independent index of stenosis severity from coronary wave-intensity analysis: results of the ADVISE (ADenosine Vasodilator Independent Stenosis Evaluation) study. J Am Coll Cardiol. 2012 Apr 10;59(15):1392-402. doi: 10.1016/j.jacc.2011.11.003. Epub 2011 Dec 7. PMID 22154731